CLINICAL TRIAL: NCT04972539
Title: A Randomized, Open, Single-dose, 2x2 Crossover Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics After Co-administration of A51R1 and A51R2 or Administration of AJU-A51 in Healthy Volunteers Under Fasting Conditions
Brief Title: Evaluation of Pharmacokinetics and Safety of AJU-A51 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20DM10202
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: AJU-A51R1 tablet(Dapagliflozin) and AJU-A51R2 tablet(Linagliptin), single dose Period 2: AJU-A51(FDC tablet, Linagliptin/Dapagliflozin), single dose
  Interventions: Drug: AJU-A51 Tab.; Drug: A51R1 Tab. and A51R2 Tab.
- Sequence B (Experimental): Period 1: AJU-A51(FDC tablet, Linagliptin/Dapagliflozin), single dose Period 2: AJU-A51R1 tablet(Dapagliflozin) and AJU-A51R2 tablet(Linagliptin), single dose
  Interventions: Drug: AJU-A51 Tab.; Drug: A51R1 Tab. and A51R2 Tab.

INTERVENTIONS:
Drug: AJU-A51 Tab. — Single oral dose AJU-A51(Dapagliflozin/Linagliptin) 10 mg / 5 mg FDC tablet
  Other Names: Test drug
Drug: A51R1 Tab. and A51R2 Tab. — Single oral dose A51R1(Dapagliflozin) 10 mg tablet and A51R2(Linagliptin) 5 mg tablet taken together
  Other Names: Reference drug

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics of AJU-A51 in healthy adults

DETAILED DESCRIPTION:
This study is to assess the safety and pharmacokinetic characteristics between co-administration of A51R1 with A51R2 and administration of AJU-A51.

This is an open-label, randomized, single-dose, 2x2 crossover study in healthy male and female subjects to assess the bioequivalence after taking the study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 19 years at the time of screening
2. Individuals who had 18.5 kg/m2 ≤ Body Mass Index(BMI) < 29.9 kg/m2 and total body weight ≥ 50 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals who were deemed to be appropriate as study subjects screening examination(laboratory tests and ECG etc.)
4. Individuals who agreed proper contraception during the study
5. Individuals who signed an informed consent form and decided to participate in the study after being fully informed of the study prior to participation

Exclusion Criteria:

1. Individuals with a medical evidence or a history of clinically significant hepatobiliary, renal, neurologic, respiratory, digestive, endocrine, blood-oncology, urinary, cardiovascular, musculoskeletal or psychiatric
2. Individuals with an active chronic or acute disease within 1 month.
3. Individuals with a medical history of gastrointestinal disease (e.g., Crohn's disease and ulcer) or gastrectomy (excluding simple appendectomy or herniotomy) that may affect drug absorption
4. Individuals with a severe allergies(except for allergic rhinitis or dermatitis)
5. Individuals with the following medical histories at screening test:

   * T1DM or diabetic ketoacidosis
   * Galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
   * Renal disorder or pancreatitis etc.
6. A history of regular alcohol consumption exceeding 21 units/week within the 3 months(1 unit = 10 g = 12.5 ml) prior to screening or individuals who cannot quit drinking from 48hr prior to the first
7. Individuals who cannot eat standard meal in institution
8. Women who are pregnant or may be pregnant
9. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
AUCt(Area Under Curve last) of AJU-A51 | predose, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72hours post-dose
  Area under the plasma concentration time curve of AJU-A51
Cmax | predose, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72hours post-dose
  The maximum concentration observed of AJU-A51 over blood sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, Principal Investigator — Chungnam National University
Locations (1):
- Jang Hee Hong, Daejeon, Korea, South Korea